CLINICAL TRIAL: NCT05569421
Title: A Phase I, Randomized, Double-blind, Single-dose, Partial-replicate, 3-way Cross-over Study to Assess the Total Systemic Exposure Bioequivalence of Budesonide, Glycopyrronium, and Formoterol Delivered by BGF MDI HFO Compared With BGF MDI HFA
Brief Title: A Study to Assess the Total Systemic Exposure Bioequivalence of of Budesonide, Glycopyrronium, and Formoterol Delivered by BGF MDI With Next-Generation Propellant Compared With BGF MDI With HFA Propellant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D5985C00004
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Bioequivalence; Propellant; Corticosteroid; Long acting muscarine agonist (LAMA); Long acting beta agonist; Lung exposure; Healthy subjects; Inhaled corticosteroid (ICS); Long-acting β2 agonist (LABA); Next generation propellant (NGP)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: BGF MDI HFO 160/7.2/4.8 μg ex-actuator (Experimental): Participants will receive Test formulation in 1 of 3 possible treatment sequences: ABB, BAB, or BBA. The reference formulation will be administered during 2 of the 3 treatment periods in order to estimate intra-subject variability.
  Interventions: Drug: Treatment A: BGF MDI HFO; Drug: Treatment B: BGF MDI HFA
- Treatment B: BGF MDI HFA 160/7.2/4.8 μg ex-actuator (Experimental): Participants will receive Reference formulation in 1 of 3 possible treatment sequences: ABB, BAB, or BBA. The reference formulation will be administered during 2 of the 3 treatment periods in order to estimate intra-subject variability.
  Interventions: Drug: Treatment A: BGF MDI HFO; Drug: Treatment B: BGF MDI HFA

INTERVENTIONS:
Drug: Treatment A: BGF MDI HFO — Participants will receive 4 oral inhalations as a single dose - test formulation; administered during 1 treatment period.
  Other Names: Budesonide/Glycopyronium/Formoterol fumarate pressurized inhalation suspension, HFO
Drug: Treatment B: BGF MDI HFA — Participants will receive 4 oral inhalations as a single dose - reference formulation; administered during 2 treatment periods.
  Other Names: Budesonide/Glycopyronium/Formoterol fumarate pressurized inhalation suspension, HFA

SUMMARY:
The study will evaluate bioequivalence, pharmacokinetics, safety, and tolerability of Budesonide, Glycopyrronium and Formoterol (BGF) metered dose inhaler (MDI) formulated with hydrofluoroolefin (HFO) [Test] and hydrofluoroalkane (HFA) [Reference] in healthy participants (male or female).

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-blind, single-dose, single-center, partial-replicate, 3 way cross-over study to assess pharmacokinetic and safety of BGF MDI when administered with different propellants, HFO (HFO-1234ze) - test and HFA (HFA-134a) - reference.

The study will comprise of:

* A screening period up to 28 days prior to first dosing;
* Three Treatment Periods: Participants will be resident at the Clinical Unit from the morning on the day before dosing with BGF MDI on Day -1 of Treatment Period 1, until 24 hours following the final dose on Day 2 of Treatment Period 3, with a washout period of 3 to 7 days between each dose; and
* Follow-up: final safety Follow-up Phone Call within 3 to 7 days after the last administration of BGF MDI in Treatment Period 3.

Each participant will receive 3 single dose treatments of BGF MDI (Treatment A: BGF MDI HFO [Test]; Treatment B: BGF MDI HFA [Reference]) following an overnight fast of at least 8 hours on Day 1 of each treatment period.

The reference formulation will be administered during 2 of the 3 treatment periods.

There will be a minimum of a 3 to 7 day washout between administration of each treatment.

Each participant will be involved in the study for approximately 55 days.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male and female subjects aged 18 to 60 years with suitable veins for cannulation or repeated venepuncture.
* Females must have a negative pregnancy test, must not be lactating
* Have a Body Mass Index (BMI) between 18 and 35 kg/m2 inclusive and weigh at least 50 kg and no more than 120 kg inclusive.
* Subjects must have a FEV1 ≥ 80% of the predicted normal value and an FEV1/FVC > 70% regarding age, height, and ethnicity.
* Subjects must demonstrate proper inhalation technique and have the ability to properly use an MDI device after training.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate.
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
* History of narrow angle glaucoma not adequately treated and/or change in vision that may be relevant.
* History of symptomatic prostatic hypertrophy or bladder neck obstruction/urinary retention that, in the opinion of the investigator, is clinically significant.
* Unresectable cancer that has not been in complete remission for at least 5 years.
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results at screening, as judged by the investigator.
* Any clinically significant abnormalities on 12-lead electrocardiogram (ECG)
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
* Subject has a positive Reverse transcriptase- Polymerase chain reaction (RT-PCR) test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
* Subject has clinical signs and symptoms consistent with SARS-CoV-2 infection, eg, fever, dry cough, dyspnea, sore throat, fatigue, or laboratory confirmed acute infection with SARS-CoV-2.
* Subject who had severe course of Corona virus disease of 2019 (COVID-19) (extracorporeal membrane oxygenation, mechanically ventilated, Intensive Care Unit stay).
* History of any respiratory disorders such as asthma, Chronic Obstructive Pulmonary Disorder (COPD), or idiopathic pulmonary fibrosis.
* Known or suspected history of alcohol or drug abuse.
* Receipt of any investigational drug within 30 days or 5 half-lives (whichever is longer) prior to randomization.
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to screening.
* Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins and minerals during the 2 weeks prior to the first administration of IMP.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* Excessive intake of caffeine-containing drinks or food. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day or would likely be unable to refrain from the use of caffeine-containing beverages during confinement.
* Subjects who have previously received BGF MDI HFO.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP and SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5985C00004&attachmentIdentifier=ebfdb998-294f-47cb-8e42-947a78a83de3&fileName=_Protocol_Main_1_EnglishD5985C00004_20_May_2024_Redacted_1.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5985C00004&attachmentIdentifier=4963e52c-eadb-4c61-bcf1-90dc09e91011&fileName=d5985c00004-CSR_Synopsis_20_May_2024_Redacted_1.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in one study center in the US.
Pre-assignment Details: The screening period was of 4 weeks. All the study assessments were performed as per the schedule of assessments. Participants who met the eligibility criteria were randomized to study intervention.
Groups:
- Treatment Sequence ABB; Treatment Sequence BAB; Treatment Sequence BBA: Participants received Test formulation in 1 of 3 possible treatment sequences: ABB, BAB, or BBA, where Treatment A: BGF MDI HFO (test), Treatment B: BGF MDI HFA (reference). The reference formulation were administered during 2 of the 3 treatment periods in order to estimate intra-subject variability.
Period: Overall Study
Arm/Group | Treatment Sequence ABB | Treatment Sequence BAB | Treatment Sequence BBA
Started | 36 | 36 | 36
Completed | 35 | 36 | 36
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The randomized analysis set consisted of all participants randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence ABB | Treatment Sequence BAB | Treatment Sequence BBA | Total
Number analyzed (Participants) | 36 | 36 | 36 | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.0 (10.0) | 35.8 (9.6) | 39.5 (11.2) | 37.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 19 | 16 | 49
  Male | 22 | 17 | 20 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 19 | 20 | 60
  Black or African American | 8 | 8 | 10 | 26
  Asian | 4 | 3 | 2 | 9
  Other | 3 | 6 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Area Under Plasma Concentration-time Curve From Zero to Infinity (AUCinf)
Description: The AUCinf of budesonide, glycopryrronium and formoterol in participants was evaluated.
Time Frame: Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
Population: The pharmacokinetic (PK) analysis set consisted of all participants in the safety analysis set for whom at least one primary PK parameter could be calculated and who had no IPDs or AEs thought to impact the analysis of the PK data. Here, N = number of participants analyzed refers to n = number analyzed for this outcome measure at specific timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*picogram/milliliter (h*pg/mL)
Groups:
- Treatment A; Treatment B (Replicate 1); Treatment B (Replicate 2): Participants received Test formulation in 1 of 3 possible treatment sequences: ABB, BAB, or BBA, where Treatment A: BGF MDI HFO (test), Treatment B: BGF MDI HFA (reference). The reference formulation were administered during 2 of the 3 treatment periods in order to estimate intra-subject variability.
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 108 | 107 | 107
hour*picogram/milliliter (h*pg/mL)
  Budesonide | 4047 (46.71) | 4112 (40.78) | 4012 (46.01)
  Glycopyronium | 85.62 (94.55) | 81.10 (78.85) | 120.9 (83.40)
  Formoterol | 124.3 (43.80) | 121.3 (41.19) | 125.0 (40.55)

2. Primary Outcome: Area Under the Plasma Concentration-curve From Zero to the Last Quantifiable Concentration (AUClast)
Description: The AUClast of budesonide, glycopryrronium and formoterol in participants was evaluated.
Time Frame: Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
Population: The PK analysis set consisted of all participants in the safety analysis set for whom at least one primary PK parameter could be calculated and who had no IPDs or AEs thought to impact the analysis of the PK data. Here, N = number of participants analyzed refers to n = number analyzed for this outcome measure at specific timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Groups:
- Treatment A; Treatment B (Replicate 1); Treatment B (Replicate 2): Participants received Test formulation in 1 of 3 possible treatment sequences: ABB, BAB, or BBA. The reference formulation were administered during 2 of the 3 treatment periods in order to estimate intra-subject variability.
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 105 | 103 | 104
h*pg/mL
  Budesonide | 3943 (47.60) | 4003 (40.66) | 3905 (46.82)
  Glycopyrronium: number analyzed (Participants) | 99 | 103 | 92
  Glycopyrronium | 52.68 (52.68) | 49.31 (84.38) | 63.29 (72.90)
  Formoterol: number analyzed (Participants) | 105 | 103 | 102
  Formoterol | 102.5 (48.47) | 100.3 (45.89) | 103.9 (42.47)

3. Primary Outcome: Maximum Observed Plasma (Peak) Drug Concentration (Cmax)
Description: The Cmax of budesonide, glycopryrronium and formoterol in participants was evaluated.
Time Frame: Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliter (pg/mL)
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 105 | 103 | 104
picograms per milliliter (pg/mL)
  Budesonide | 1124 (65.67) | 1143 (60.79) | 1146 (65.91)
  Glycopyrronium: number analyzed (Participants) | 100 | 103 | 93
  Glycopyrronium | 17.09 (90.52) | 20.41 (87.46) | 19.70 (87.52)
  Formoterol: number analyzed (Participants) | 105 | 103 | 103
  Formoterol | 23.48 (60.12) | 24.54 (62.22) | 26.12 (54.39)

4. Secondary Outcome: Time to Reach Peak or Maximum Observed Concentration or Response Following Drug Administration (Tmax)
Description: The tmax of budesonide, glycopryrronium and formoterol in participants was evaluated.
Time Frame: Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 105 | 103 | 104
Hours
  Budesonide | 0.35 [0.08 to 2.00] | 0.33 [0.08 to 2.02] | 0.33 [0.07 to 2.05]
  Glycopyrronium: number analyzed (Participants) | 100 | 103 | 93
  Glycopyrronium | 0.03 [0.02 to 4.13] | 0.03 [0.03 to 2.02] | 0.03 [0.02 to 4.02]
  Formoterol: number analyzed (Participants) | 105 | 103 | 103
  Formoterol | 0.08 [0.03 to 4.02] | 0.08 [0.03 to 2.03] | 0.08 [0.03 to 2.12]

5. Secondary Outcome: Terminal Rate Constant, Estimated by Log-linear Least Squares Regression of the Terminal Part of the Concentration-time Curve (λz)
Description: The λz of budesonide, glycopryrronium and formoterol in participants was evaluated.
Time Frame: Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 105 | 103 | 104
1/hour
  Budesonide | 0.1508 (25.19) | 0.1538 (25.24) | 0.1500 (24.99)
  Glycopyrronium: number analyzed (Participants) | 93 | 95 | 78
  Glycopyrronium | 0.05906 (97.13) | 0.06010 (92.16) | 0.03853 (100.5)
  Formoterol: number analyzed (Participants) | 103 | 102 | 102
  Formoterol | 0.08911 (36.39) | 0.08926 (36.50) | 0.08625 (39.39)

6. Secondary Outcome: Half-life Associated With Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t½λz)
Description: The t½λz of budesonide, glycopryrronium and formoterol in participants was evaluated.
Time Frame: Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 105 | 103 | 104
Hours
  Budesonide | 4.596 (25.19) | 4.506 (25.24) | 4.622 (24.99)
  Glycopyrronium: number analyzed (Participants) | 93 | 95 | 78
  Glycopyrronium | 11.74 (97.13) | 11.53 (92.16) | 17.99 (100.5)
  Formoterol: number analyzed (Participants) | 103 | 102 | 102
  Formoterol | 7.779 (36.39) | 7.766 (36.50) | 8.037 (39.39)

7. Secondary Outcome: Mean Residence Time of the Unchanged Drug in the Systemic Circulation From Zero to Infinity (MRTinf)
Description: The MRTinf of budesonide, glycopryrronium and formoterol in participants was evaluated.
Time Frame: Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 105 | 103 | 104
Hours
  Budesonide | 4.855 (21.37) | 4.893 (24.30) | 4.924 (19.98)
  Glycopyrronium: number analyzed (Participants) | 93 | 95 | 78
  Glycopyrronium | 16.02 (93.66) | 15.56 (86.14) | 24.50 (96.84)
  Formoterol: number analyzed (Participants) | 103 | 102 | 102
  Formoterol | 10.48 (29.28) | 10.38 (30.42) | 10.62 (33.34)

8. Secondary Outcome: Apparent Total Body Clearance of Drug From Plasma After Extravascular Administration (CL/F)
Description: The CL/F of budesonide, glycopryrronium and formoterol in participants was evaluated.
Time Frame: Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour (L/h)
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 105 | 103 | 104
Liters/hour (L/h)
  Budesonide | 158.2 (46.71) | 155.6 (40.78) | 159.5 (46.01)
  Glycopyrronium: number analyzed (Participants) | 93 | 95 | 78
  Glycopyrronium | 336.4 (94.55) | 355.1 (78.85) | 238.2 (83.40)
  Formoterol: number analyzed (Participants) | 103 | 102 | 102
  Formoterol | 154.5 (43.80) | 158.2 (41.19) | 153.6 (40.55)

9. Secondary Outcome: Volume of Distribution (Apparent) at Steady State Following Extravascular Administration (Based on Terminal Phase) (Vz/F)
Description: The Vz/F of budesonide, glycopryrronium and formoterol in participants was evaluated.
Time Frame: Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 105 | 103 | 104
Liters (L)
  Budesonide | 1049 (47.84) | 1012 (39.18) | 1064 (45.06)
  Glycopyrronium: number analyzed (Participants) | 93 | 95 | 78
  Glycopyrronium | 5695 (43.16) | 5908 (46.44) | 6182 (44.59)
  Formoterol: number analyzed (Participants) | 103 | 102 | 102
  Formoterol | 1734 (32.78) | 1773 (33.69) | 1782 (36.52)

10. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: The safety and tolerability of single doses of BGF MDI HFO and BGF MDI HFA was evaluated in healthy participants.
Time Frame: From Screening up to Follow-up (3 to 7 days post final dose) [approximately 55 days]
Population: The safety analysis set included all participants who received at least one inhalation of any BGF MDI.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
Number analyzed (Participants) | 108 | 107 | 107
Participants
  Any AEs | 16 | 21 | 9
  Any SAE | 0 | 0 | 0
  Any SAE with outcome of death | 0 | 0 | 0
  Any AE leading to discontinuation of Investigational Product (IP) | 0 | 0 | 0
  Any possibly related AE | 10 | 12 | 4
  Any possibly related SAE | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Screening up to Follow-up Phone call (3 to 7 days post final dose) [approximately 55 days]
Arm/Group | Treatment A | Treatment B (Replicate 1) | Treatment B (Replicate 2)
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/107 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/107 | 0/107
Other Adverse Events (participants affected / at risk) | 16/108 | 21/107 | 9/107
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=108) | Treatment B (Replicate 1) (N=107) | Treatment B (Replicate 2) (N=107)
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 1
Headache (Nervous system disorders) | 4 | 8 | 1
Hypoaesthesia eye (Eye disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Salivary gland mucocoele (Gastrointestinal disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Catheter site bruise (General disorders) | 2 | 1 | 1
Catheter site pain (General disorders) | 0 | 1 | 2
Catheter site related reaction (General disorders) | 0 | 1 | 0
Catheter site swelling (General disorders) | 0 | 0 | 2
Chest discomfort (General disorders) | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Thirst (General disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This confidential document is the property of AstraZeneca AB. No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca AB. Access to this document must be restricted to relevant parties.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT05569421/Prot_SAP_000.pdf